CLINICAL TRIAL: NCT00625807
Title: Exploratory Analysis of the Relaxation Response (RR) and Mindfulness Based Stress Reduction (MBSR) for Stress Reduction
Brief Title: Comparison of Two Behavioral Treatments for Stress Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Sara W Lazar, Associate Research Scientist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21AT003425-01A2 (NIH); R21AT003425-01A2 (NIH); SL1
Record Dates: First submitted 2008-02-26; First posted 2008-02-28 (Estimated); Results first posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-07

CONDITIONS: Stress
Keywords: Stress; meditation; stress reduction; fMRI; behavioral
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Program A - Relaxation Response (RR) (Active Comparator): One of the 2 stress reduction courses
  Interventions: Behavioral: RR
- Program B - Mindfullness-based stress reduction (MBSR) (Active Comparator): One of the 2 stress reduction courses
  Interventions: Behavioral: MBSR

INTERVENTIONS:
Behavioral: RR — A well-validated 8 week stress reduction course. Classes meet once a week for 1.5 hours. Participants will be asked to perform stress reduction techniques each night for 20 minutes throughout the entire 8-week course. Stress reduction techniques use meditative techniques that focus primarily on inducing relaxation
  Arms: Program A - Relaxation Response (RR)
Behavioral: MBSR — A well-validated 8 week stress reduction course. Classes meet once a week for 1.5 hours. Participants will be asked to perform stress reduction techniques each night for 20 minutes throughout the entire 8-week course. Stress reduction techniques use meditative techniques that focus primarily on inducing mindfulness
  Arms: Program B - Mindfullness-based stress reduction (MBSR)

SUMMARY:
Currently there are 2 popular stress reduction courses that are widely used in the US. Although they use somewhat similar techniques, it is currently unknown whether or not they work the same way, or if they are similarly effective at reducing stress. The study will directly compare these 2 courses. Participants will undergo approximately 4-5 hours of testing before and after each 8-week course.

ELIGIBILITY:
Inclusion Criteria:

* 25 to 60 years old
* Good general health
* Able to attend all 8 sessions of the course and practice the techniques each night for 25 minutes

Exclusion Criteria:

* Psychiatric medications
* Significant medical or psychological illness
* Metalic implants (such as a pacemaker or artificial joints) that are not MRI compatible.
* Claustrophobia
* Pregnancy
* Previous head trauma or neurological disorder
* Previous experience with yoga or meditation

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2008-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Lazar, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Relaxation Response (RR): One of the 2 stress reduction courses
  A well-validated 8 week stress reduction course. Classes meet once a week for 1.5 hours. Participants will be asked to perform stress reduction techniques each night for 20 minutes throughout the entire 8-week course. Stress reduction techniques use meditative techniques that focus primarily on inducing relaxation
- Mindfulness Based Stress Reduction (MBSR): One of the 2 stress reduction courses
  A well-validated 8 week stress reduction course. Classes meet once a week for 1.5 hours. Participants will be asked to perform stress reduction techniques each night for 20 minutes throughout the entire 8-week course. Stress reduction techniques use meditative techniques that focus primarily on inducing mindfulness
Period: Overall Study
Arm/Group | Relaxation Response (RR) | Mindfulness Based Stress Reduction (MBSR)
Started | 22 | 28
Completed | 20 | 20
Not Completed | 2 | 8
Not completed — schedule conflict | 2 | 8

BASELINE CHARACTERISTICS:
Groups:
- Relaxation Response: One of the 2 stress reduction courses
  Relaxation Response: A well-validated 8 week stress reduction course. Participants will be asked to perform stress reduction techniques from the Relaxation Response Program each night for 20 minutes throughout the entire 8-week course
- MBSR: One of the 2 stress reduction courses
  MBSR: A well-validated 8 week stress reduction course. Classes meet once a week from 5-8:30 PM. Participants will be asked to perform stress reduction techniques from the MBSR program each night for 20 minutes throughout the entire 8-week course
- Total: Total of all reporting groups
Arm/Group | Relaxation Response | MBSR | Total
Number analyzed (Participants) | 22 | 28 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (8.7) | 37 (4.7) | 37.9 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 18 | 33
  Male | 7 | 10 | 17

OUTCOME MEASURES:

1. Primary Outcome: Brain Activity (fMRI) During the Body Scan Meditation
Description: Seed based functional connectivity analysis was performed using the Connectivity Toolbox (CONN) implemented within the Statistical Parametric Mapping program (SPM8; Welcome Department of Cognitive Neurology). Our seeds were located in the right inferior frontal gyrus pars opercularis (MNI coordinates: 54, 14, 16) and the dorsal anterior insula (MNI coordinates: 32, 20, 0). Note - MRI data from some subjects was either missing, not collected, or corrupted, and so the analyses were performed on just the subject of subjects who had complete datasets. This assessment reflects the total number of voxels per group.
Time Frame: Week 8
Measure: Number; unit: voxels
Arm/Group | Relaxation Response (RR) | Mindfulness Based Stress Reduction (MBSR)
Number analyzed (Participants) | 16 | 18
voxels | 74 | 82

2. Primary Outcome: Five Facet Mindfulness Questionnaire
Description: The Five Facet Mindfulness Questionnaire (FFMQ) has been developed as a reliable and valid comprehensive instrument for assessing different aspects of mindfulness in community samples. Scores range from 39-195 with higher scores meaning more mindfulness.
Time Frame: Pre, 8 weeks
Population: Individuals who completed at least one measure at post
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Relaxation Response: One of the 2 stress reduction courses
  A well-validated 8 week stress reduction course. Participants were asked to perform stress reduction techniques each night for 20 minutes throughout the entire 8-week course. Meditation techniques focused on developing relaxation
- MBSR: One of the 2 stress reduction courses
  A well-validated 8 week stress reduction course. Participants were asked to perform stress reduction techniques each night for 20 minutes throughout the entire 8-week course. Meditation techniques focused on developing mindfulness
Arm/Group | Relaxation Response | MBSR
Number analyzed (Participants) | 20 | 20
units on a scale
  Pre | 130.8 (17.7) | 125.3 (17.7)
  week 8 | 144.2 (20.6) | 139.1 (21.1)
Statistical Analysis 1: Comparison: Relaxation Response vs MBSR; ANOVA for group by time interaction; Test type: Other; p > 0.1, ANOVA — Cohen's d = 0.5

3. Primary Outcome: Perceived Stress Scale
Description: The PSS is brief, validated and widely used psychological instrument for assessing a subject's perception of stress change. Scores range from 0-40 with higher scores meaning more stress
Time Frame: Pre, 8 weeks
Population: Individuals who completed at least one measure at post
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Relaxation Response | MBSR
Number analyzed (Participants) | 20 | 20
units on a scale
  Pre | 14.1 (6.6) | 18.4 (6.7)
  week 8 | 11.3 (5.5) | 12.3 (5.3)
Statistical Analysis 1: Comparison: Relaxation Response vs MBSR; Test type: Other; p = 0.103, ANOVA

4. Primary Outcome: Penn State Worry Questionnaire
Description: The Penn State Worry Questionnaire (PSWQ) is a standard self-report questionnaire that is designed to assess symptoms of General Anxiety Disorder. scores range from 16-80 with higher scores meaning more stress.
Time Frame: Pre, 8 weeks
Population: Individuals who completed at least one measure at post
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Relaxation Response | MBSR
Number analyzed (Participants) | 19 | 18
units on a scale
  Pre | 42.6 (11.9) | 50.5 (13.1)
  week 8 | 37.7 (10.1) | 44.3 (12.0)
Statistical Analysis 1: Comparison: Relaxation Response; within group change pre to week 8; Test type: Other; p = .022, t-test, 2 sided
Statistical Analysis 2: Comparison: MBSR; Test type: Other — within group change from pre to week 8; p < .001, t-test, 2 sided

5. Primary Outcome: Anxiety Severity Index
Description: the Anxiety Sensitivity Index (ASI) is a measure of individuals discomfort with a variety of sensations associated with anxiety and panic and tends to be substantially higher in those with panic disorder (and attacks) than in those with General Anxiety Disorder. Scores range from 0 - 64. Lower scores mean lower anxiety.
Time Frame: Pre, 8 weeks
Population: Individuals who completed at least one measure at post
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Relaxation Response | MBSR
Number analyzed (Participants) | 18 | 19
units on a scale
  Pre | 29.8 (7.3) | 31.9 (9.4)
  week 8 | 25.4 (5.7) | 30.9 (8.6)
Statistical Analysis 1: Comparison: Relaxation Response; within group change from pre to week 8; Test type: Other; p = .015, t-test, 2 sided
Statistical Analysis 2: Comparison: MBSR; within group change from pre to week 8; Test type: Other; p = .53, t-test, 2 sided

6. Secondary Outcome: Self Compassion
Description: This scale assesses one's ability to be forgiving and kind to oneself in difficult circumstances. Scores range from 1-5. Higher scores mean more self compassion.
Time Frame: Pre, week 8
Population: individuals who completed the measure at week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Relaxation Response | MBSR
Number analyzed (Participants) | 20 | 20
units on a scale
  pre | 2.9 (.67) | 3.1 (.6)
  week 8 | 3.2 (.72) | 3.6 (.7)
Statistical Analysis 1: Comparison: Relaxation Response; within group change from pre to week 8; Test type: Other; p = .06, t-test, 2 sided
Statistical Analysis 2: Comparison: MBSR; within group change from pre to post; Test type: Other; p < .001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 2 months
Description: Participants were given a daily log in which to record their daily meditation practice, overall stress levels, and any information about their practice or unusual occurances that they wished to share with the study team. Any individual who missed a class or dropped out of the study were contacted to determine the reason.
Groups:
- Relaxation Response: One of the 2 stress reduction courses
  Program A: A well-validated 8 week stress reduction course. Classes meet once a week from 5-8:30 PM. Participants will be asked to perform stress reduction techniques each night for 20 minutes throughout the entire 8-week course
- MBSR: One of the 2 stress reduction courses
  Program B: A well-validated 8 week stress reduction course. Classes meet once a week from 5-8:30 PM. Participants will be asked to perform stress reduction techniques each night for 20 minutes throughout the entire 8-week course
Arm/Group | Relaxation Response | MBSR
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/28
Other Adverse Events (participants affected / at risk) | 0/22 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes